CLINICAL TRIAL: NCT00846287
Title: Assessment of Arformoterol for COPD Using Hyperpolarized 3He MRI
Brief Title: Assessment of Arformoterol for Chronic Obstructive Pulmonary Disease (COPD) Using Hyperpolarized 3He MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Mitchell Albert, Director of Advanced MRI Center, UMASS Medical Sch, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Docket # 12830
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; aformoterol; Helium; Hyperpolarized helium; Hyperpolarized Noble Gas; MRI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Sodium Chloride; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Subjects (Active Comparator): Patients will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. The first three bags will be administered with a break between each of five to ten minutes. Then the drug aformoterol will be administered and an hour will pass. BROVANA (arformoterol tartrate) Inhalation Solution is supplied as 2 mL of arformoterol tartrate solution packaged in 2.1 mL unit-dose, low-density polyethylene (LDPE) unit-dose vials. Each unit-dose vial contains 15 mcg of arformoterol (equivalent to 22 mcg of arformoterol tartrate) in a sterile, isotonic saline solution, pH-adjusted to 5.0 with citric acid and sodium citrate. After administration of the drug, three additional bags of hyperpolarized helium-3 will be administered, again with five to ten minutes between each bag.
  Interventions: Drug: Hyperpolarized Helium-3; Drug: Aformoterol
- Saline (Placebo Comparator): Patients will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. The first three bags will be administered with a break between each of five to ten minutes. Then the placebo (nebulized saline solution) will be administered (2.1 mL). After administration of the placebo, three additional bags of hyperpolarized helium-3 will be administered, again with five to ten minutes between each bag.
  Interventions: Drug: Hyperpolarized Helium-3; Drug: Placebo

INTERVENTIONS:
Drug: Hyperpolarized Helium-3 — Patients will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. The first three bags will be administered with a break between each of five to ten minutes. Then the intervention (drug or placebo) will be administered and an hour will pass. Then three additional bags will be administered, again with five to ten minutes between each bag.
  Other Names: HP 3He
Drug: Placebo — Subject will inhale a placebo (nebulized saline) with no drug.
  Other Names: Saline
  Arms: Saline
Drug: Aformoterol — Subjects will receive the drug arformoterol prior to scanning
  Other Names: Brovana
  Arms: Drug Subjects

SUMMARY:
The purpose of this study is to determine efficacy of MR imaging with hyperpolarized helium-3 gas in COPD patients both before and after treatment.

DETAILED DESCRIPTION:
Hyperpolarized Helium Lung imaging has already been tested and proven to be scientifically possible in patients with a number of pulmonary disorders. However there is limited data on the sensitivity of this imaging technique, which would be essential for clinical use. This study is a double blinded study with two cohorts, each cohort being made up of patients with confirmed diagnosis of COPD. One group will receive a placebo while the other will receive treatment. A comparison of the data will resume once twenty patients have been consented and completed the study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female and are 50 years or older
* Consent from the patient
* Have been diagnosed with COPD
* Must be able to hold their breath for up to 12 seconds
* Must have a baseline FEV1 ≤ 80% of predicted but FEV1 > 0.70 L
* Must have a smoking history of 15 or more packs per year
* Must have a breathlessness severity of ≥ 2 on the Medical Research Council dyspnea scale
* Must be able to safely discontinue their respiratory medications for at least 12 hours.

Exclusion Criteria:

* Have any contraindications to an MR exam such as a pace-maker, metallic cardiac valves, magnetic material (i.e., surgical clips) implanted electronic infusion pumps or any other conditions that would preclude proximity to a strong magnetic field
* Are undergoing the MR exam in an emergency situation
* Are pregnant or become pregnant at any point within the study time.
* People with psychiatric disorders will be excluded from the study.
* Are claustrophobic and can not tolerate the imaging.
* Uses supplemental oxygen
* Have life-threatening or unstable respiratory status within 30 days before screening
* Have a diagnosis of asthma and/or any chronic respiratory disease other than COPD
* Have a lung resection greater than 1 full lobe
* Have coronary artery disease or congestive heart failure
* Are allergic to Arformoterol or similarly related drugs.
* Are taking any of the drugs listed in the risks section and are unable to stop taking them.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Albert, Ph.D., Principal Investigator — UMASS Medical School
Locations (1):
- UMASS Medical School Advanced MRI Center, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with moderate to severe COPD were recruited and enrolled from the UMass Lung and Allergy Center from November 2008 to April 2011.
Groups:
- Active Comparator: Saline: Subjects (n=10) will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of hyperpolarized Helium-3 gas and 667mL of Nitrogen. The first three bags will be administered with a break between each of five to ten minutes. Then the placebo will be administered and an hour will pass. The placebo consists of a nebulized saline solution (2.1 mL). After administration of the placebo, three additional bags of hyperpolarized helium-3 will be administered, again with five to ten minutes between each bag.
- Active Comparator: Drug Subjects: Subjects (n=10) will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of hyperpolarized Helium-3 gas and 667mL of Nitrogen. The first three bags will be administered with a break between each of five to ten minutes. Then the drug aformoterol will be administered and an hour will pass. BROVANA (arformoterol tartrate) Inhalation Solution is supplied as 2 mL of arformoterol tartrate solution packaged in 2.1 mL unit-dose, low-density polyethylene (LDPE) unit-dose vials. Each unit-dose vial contains 15 mcg of arformoterol (equivalent to 22 mcg of arformoterol tartrate) in a sterile, isotonic saline solution, pH-adjusted to 5.0 with citric acid and sodium citrate. After administration of the drug, three additional bags of hyperpolarized helium-3 will be administered, again with five to ten minutes between each bag.
Period: Overall Study
Arm/Group | Active Comparator: Saline | Active Comparator: Drug Subjects
Started | 16 | 15
Completed | 6 | 10
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Saline: Subjects will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of hyperpolarized Helium-3 gas and 667mL of Nitrogen. The first three bags will be administered with a break between each of five to ten minutes. Then the placebo will be administered and an hour will pass. The placebo consists of a nebulized saline solution (2.1 mL). After administration of the placebo, three additional bags of hyperpolarized helium-3 will be administered, again with five to ten minutes between each bag.
- Drug Subjects: Subjects will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of hyperpolarized Helium-3 gas and 667mL of Nitrogen. The first three bags will be administered with a break between each of five to ten minutes. Then the drug aformoterol will be administered and an hour will pass. BROVANA (arformoterol tartrate) Inhalation Solution is supplied as 2 mL of arformoterol tartrate solution packaged in 2.1 mL unit-dose, low-density polyethylene (LDPE) unit-dose vials. Each unit-dose vial contains 15 mcg of arformoterol (equivalent to 22 mcg of arformoterol tartrate) in a sterile, isotonic saline solution, pH-adjusted to 5.0 with citric acid and sodium citrate. After administration of the drug, three additional bags of hyperpolarized helium-3 will be administered, again with five to ten minutes between each bag.
- Total: Total of all reporting groups
Arm/Group | Saline | Drug Subjects | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 8 | 8 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (7) | 68 (11) | 66 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Ventilation Volume
Description: Subjects had hyperpolarized helium-3 MR scans completed before administration of an intervention and 2 hours after administration. These images were compared as described:
  The change in the total ventilation volume (Litres) measured in the hyperpolarized helium-3 MR image from pre-nebulizer inhalation to post-nebulizer inhalation.
Time Frame: 2 hours
Population: Analysis per protocol.
Measure: Mean (Standard Deviation); unit: Litres
Groups:
- Placebo Subjects: Subjects will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of hyperpolarized Helium-3 gas and 667mL of Nitrogen. The first three bags will be administered with a break between each of five to ten minutes. Then the placebo will be administered and an hour will pass. The placebo consists of a nebulized saline solution (2.1 mL). After administration of the placebo, three additional bags of hyperpolarized helium-3 will be administered, again with five to ten minutes between each bag
- Brovana Subjects: Subjects (n=10) will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of hyperpolarized Helium-3 gas and 667mL of Nitrogen. The first three bags will be administered with a break between each of five to ten minutes. Then the drug aformoterol will be administered and an hour will pass. BROVANA (arformoterol tartrate) Inhalation Solution is supplied as 2 mL of arformoterol tartrate solution packaged in 2.1 mL unit-dose, low-density polyethylene (LDPE) unit-dose vials. Each unit-dose vial contains 15 mcg of arformoterol (equivalent to 22 mcg of arformoterol tartrate) in a sterile, isotonic saline solution, pH-adjusted to 5.0 with citric acid and sodium citrate. After administration of the drug, three additional bags of hyperpolarized helium-3 will be administered, again with five to ten minutes between each bag.
Arm/Group | Placebo Subjects | Brovana Subjects
Number analyzed (Participants) | 6 | 10
Litres | 0.154317 (0.512) | -0.13687 (0.306)

2. Secondary Outcome: Change in FEV1
Description: Spirometry was taken which measures FEV1 (in Litres), before administration of an intervention and again 2 hours after administration of an intervention. The change in FEV1 (Litres) from pre-nebulizer inhalation to post-nebulizer inhalation was compared.
Time Frame: 2 hours
Population: As per protocol
Measure: Median (Standard Deviation); unit: Litres
Arm/Group | Placebo Subjects | Brovana Subjects
Number analyzed (Participants) | 6 | 10
Litres | -0.12 (0.25) | 0.16 (0.26)

ADVERSE EVENTS:
Arm/Group | Saline | Drug Subjects
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less